CLINICAL TRIAL: NCT00057564
Title: A Multicenter, Randomized, Parallel-group , Double Blind, Placebo-controlled Study of Combination Thalidomide Plus Dexamethasone Therapy vs. Dexamethasone Therapy Alone as Induction Therapy for Previously Untreated Subjects With Multiple Myeloma
Brief Title: A Study of Combination Thalidomide Plus Dexamethasone Therapy vs. Dexamethasone Therapy Alone in Previously Untreated Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THAL-MM-003
Record Dates: First submitted 2003-04-04; First posted 2003-04-07 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Multiple Myeloma
Keywords: Newly Diagnosed Multiple Myeloma; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Thalidomide & Dexamethasone) (Experimental): Thalidomide 50mg/day + Dexamethasone 40mg
  Interventions: Drug: A (Thalidomide + Dexamethasone)
- B (Dexamethasone and placebo) (Placebo Comparator): Dexamethasone and placebo
  Interventions: Drug: B (Placebo + Dexamethasone)

INTERVENTIONS:
Drug: A (Thalidomide + Dexamethasone) — Thalidomide 50mg/day + Dexamethasone 40mg
  Other Names: Thalidomide
  Arms: A (Thalidomide & Dexamethasone)
Drug: B (Placebo + Dexamethasone) — Placebo + Dexamethasone 40mg
  Other Names: Dexamethasone; placebo
  Arms: B (Dexamethasone and placebo)

SUMMARY:
To compare the efficacy of combination oral thalidomide plus oral dexamethasone treatment to that of oral dexamethasone-alone treatments as induction (first-line) therapy for subjects with active multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

* Active Multiple Myeloma Stage II or III Durie Salmon
* Measurable levels of myeloma paraprotein in serum (≥1.0g/dL) or urine (≥ 0.2g excreted in a 24-hour collection sample)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, 2
* Women of child bearing potential must agree to abstain for heterosexual intercourse or use 2 methods of contraception, one effective (for example hormonal or tubal ligation) and one barrier (for example latex condom, diaphragm)
* Males must agree to use barrier contraception (latex condoms) when engaging in reproductive activity

Exclusion Criteria:

* Pregnant or lactating females
* Peripheral neuropathy ≥ to grade 2 of the NCI CTC.
* Prior history of malignancy unless subject has been free of disease for ≥ 3 years
* Lab abnormality: Absolute neutrophil count (ANC) <1,000 cells/mm^3 (1.0 x 10^9/L)
* Lab abnormality: Platelet count <50,000/mm^3 (50.0 x 10^9/L)
* Lab abnormality: Serum creatinine >3.0 mg/dL (265 µmol/L)
* Lab abnormality: Serum glutamic oxaloacetic transaminase (SGOT) /Aspartate aminotransferase (AST) or Serum glutamic pyruvic transaminase (SGPT)/Alanine transaminase (ALT) >3.0 x upper limit of normal (ULN)
* Lab abnormality: Serum total bilirubin > 2.0 mg/dL (34 µmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2003-02; Primary Completion 2006-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Time to tumor progression (TTP) | Up to 3 years
  Time to tumor progression (TTP)

SECONDARY OUTCOMES:
Number of patients who survived | Up to 3 years
  Number of patients who survived
Time to first symptomatic skeletal-related event (SRE)(clinical need for radiation therapy or surgery to bone) | Up to 3 years
  Time to first symptomatic skeletal-related event (SRE)(clinical need for radiation therapy or surgery to bone)
Myeloma response rate | Up to 3 years
  Myeloma response determination criteria developed by Bladé et al 1998
Number of participants with adverse events | Up to 3 years
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Director — Celgene Corporation
Locations (98):
- United States (26):
  - Clinical Research Consultants, Inc., Hoover, Alabama
  - Arizona Clinical Research Center, Tucson, Arizona
  - UCLA School of Medicine, Los Angeles, California
  - James Berenson, West Hollywood, California
  - Mayo Clinic, Jacksonville, Florida
  - Melbourne Internal Medicine Associates Oncology, Melbourne, Florida
  - Jackson Memorial Hospital and Clinics, Miami, Florida
  - University of Miami Miller School/Jackson Memorial Hospital, Miami, Florida
  - University of Miami, Miami, Florida
  - Oncology Hematology Group of South Florida, Miami, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Southern Illinois Hematology /Oncology, Centralia, Illinois
  - Rush Cancer Institute Section of Hematology, Chicago, Illinois
  - University of Iowa Hospital of Clinic, Iowa City, Iowa
  - Ocshner Clinic Foundation, New Orleans, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Hackensack University Hospital, Hackensack, New Jersey
  - SUNY Upstate Medical University, Syracuse, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic- Taussig Cancer Center, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - South Carolina Oncology Group, West Columbia, South Carolina
  - The Family Centre, PLLC, Collierville, Tennessee
  - East Tennessee Oncology/Hematology Associates, Knoxville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - Royal Brisbane Hospital, Herston, Queensland
  - Haematology Princess Alexandra Hospital, Woolloongabba, Queensland
  - Frankston Hospital, Frankston, Victoria
  - Peter MacCallum Cancer Institute, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Bone Marrow Transplant Service Dept of Clinical Haematology and Medical Oncology, Parkville, Victoria
- Belgium (3):
  - Institut Jules Bordet Dep't of Clinical Haematology, Brussels
  - Dept. Of Haematology Academisch Ziekenhuis VUB, Brussels
  - University Hospital Ghent Dep't of Haematology, Ghent
- Bulgaria (3):
  - UMHAT Alexandrovska, Alexandrovska
  - National Center of Haematology and Transfusiology, Sofia
  - Military Medical Academy, Sofia
- Canada (6):
  - Dalhousie University, Halifax, Nova Scotia
  - Princess Margaret Hospital, Toronto, Ontario
  - University Health Network Princess Margaret Hospital, Toronto, Ontario
  - Centre Hopitalier Universitaire de Sherbrooke Hospital Fleurimont, Fleurimont, Quebec
  - McGill University, Montreal, Quebec
  - Saskatoon Cancer Centre University of Saskatoon, Saskatoon, Saskatchewan
- Universitaetsklinikum Dusseldorf Klinik fuer Haematologie, Düsseldorf, Germany
- Hungary (2):
  - St. Laszlo Hoszpital, Budapest
  - Petz Aladar County Hospital, Győr
- Ireland (2):
  - MidWestern Regional Hospital Haematology Dpt., Dooradoyle, Limerick
  - Hope Directorate Dep't. Haematology St. James's Hospital, Dublin
- Israel (4):
  - Hadassah University Hospital Hematology Dep't, ‘En Kerem, Jerusalem
  - Rambam Medical Center Dep't. Of Hematology, Haifa
  - Tel Aviv Sourasky Medical Center Hematology Institute, Tel Aviv
  - Director of Hematology Division BMT and CBB The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (7):
  - Universita di Bari Dipartimento di Scienze Umana Sezione de Medicina Interna e Oncologia Medica Policlinico, Bari
  - Istituto di Ematologia e Oncologia Medica "L. e. A. Seragnoli", Bologna
  - Azienda Ospedaliera San Martino, Genova
  - Ospedale Niguarda Ca Granda, Milan
  - Policlinico San Matteo, Pavia
  - Università La Sapienza Dipartimento di Biotecnologie Cellulari ed Ematologia, Roma
  - Clinica Ematologica Policlinico Universitario, Udine
- Poland (6):
  - Medical Academy of Bialystok, Bialystok
  - Institute of Internal Diseases University of Medicine, Gdansk
  - Jagiellonian University Collegium Medicum Department of Hematology, Krakow
  - Medical University of Lodz, Lodz
  - Private Medical Practice Centre of Clinical Laboratory of Densitometry At 'Officers of Professors', Lublin
  - Medical University of Warsaw Dep't of Hematology, Oncology and Internal Diseases, Warsaw
- Russia (12):
  - Chelyabinsk Regional Clinical Hospital Hematology Dpt, Chelyabinsk
  - Republican Clinical Hospital #1 Hematology Dpt., Izhevsk
  - Burdenko Central Military Clinical Hospital Hematology Center, Moscow
  - Russian Academy of Medical Sciences Scientific Center of Hematology, Moscow
  - Novosibirsk State Regional Clinical Hospital Hematology Centre, Novosibirsk
  - Research Institute of Hematology and Blood Transfusion,Clinical Department of Hematology with Bone Marrow Transplantation Unit, Saint Petersburg
  - St. Petersburg Pavlov State Medical University Bone Marrow Transplantation Clinic, Saint Petersburg
  - Clinical Hospital #31 Dpt of Bone Marrow Transplantation and Chemotherapy of Patients with Myeloproliferative Disorders, Saint Petersburg
  - Samara Regional Clinical Hospital Dep't. of Hematology and Bone Marrow Transplantation, Samara
  - Blokhin Cancer Research Center Dpt of Myeloproliferative Disorders Chemotherapy, Shosse
  - Nizhny Novgorod Clinical Hospital, Veliky Novgorod
  - Ekaterinburg 1st Regional Clinical Hospital Regional Hematology Centre, Yekaterinburg
- Spain (6):
  - Hospital Clinic, Barcelona
  - Hospital Universitario de la Princessa, Madrid
  - Hospital Doce de Octubre, Madrid
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
- Universitatsspital Zurich, Zurich, Switzerland
- Ukraine (11):
  - Cherkassy Regional Oncology Center, Cherkassy
  - Dnepropetrovsk City Clinical Hospital #4 Regional Hematology Centre, Dnipro
  - Ivano-Frankovsk Regional Clinical Hospital - Hospital Therapy Department, Ivano-Frankivsk
  - Kharkov Regional Clinical Oncology Center Dep't of Oncology and Pediatric Oncology, Kharkiv
  - Kiev Institute of Oncology of the UAMS Systemic Malignancies Department, Kiev
  - Kiev Bone Marrow Transplantation Center Bone Marrow Transplantation Department, Kiev
  - Institute of Hematology and Transfusiology of the UAMS Department of Blood Diseases with Clinical Biochemistry Group, Kiev
  - Institute of Blood Pathology and Transfusion Medicine of the UAMS, Lviv
  - Odessa Regional Clinical Hospital Hematology Dep't, Odesa
  - Zaporozhje Regional Clinical Hospital Hematology Dpt, Zaporizhzhya
  - Zhitomir Regional Clinical Hospital Hematology Centre, Zhytomyr
- United Kingdom (2):
  - Belfast City Hospital Haematology Dpt., Belfast
  - Guys Hospital, London

REFERENCES:
- [Result] Rajkumar SV, Rosinol L, Hussein M, Catalano J, Jedrzejczak W, Lucy L, Olesnyckyj M, Yu Z, Knight R, Zeldis JB, Blade J. Multicenter, randomized, double-blind, placebo-controlled study of thalidomide plus dexamethasone compared with dexamethasone as initial therapy for newly diagnosed multiple myeloma. J Clin Oncol. 2008 May 1;26(13):2171-7. doi: 10.1200/JCO.2007.14.1853. Epub 2008 Mar 24. PMID 18362366